CLINICAL TRIAL: NCT00940563
Title: STI571 (Imatinib) in KIT-expressing Gastrointestinal Stromal Tumors (GIST): a Prospective, Open-label, Multicenter Study on Best Clinical Use in the Advanced Disease.
Brief Title: A Prospective, Multicenter Study on Best Clinical Use of Imatinib in the Advanced Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BIT03; NCT00942279 (obsolete NCT alias)
Record Dates: First submitted 2009-06-26; First posted 2009-07-16 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Advanced Gastrointestinal Stromal Tumors
Keywords: GIST; imatinib; advanced GIST
MeSH Terms: interventions — Imatinib Mesylate

ARMS (1):
- Imatinib (Experimental)
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib

SUMMARY:
Open-label, multicenter study of imatinib (400mg/die p.o.)in patients with advanced gastrointestinal stromal tumors. Patients will be treated for up to 12 months. Data regarding its best clinical use in terms of tumor response, survival, tolerability and safety profile will be prospectively collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Histologically documented diagnosis of GIST, unresectable and/or metastatic and therefore incurable with any conventional multimodality approach.
3. Immunohistochemical documentation of c-kit (CD117) expression by tumor, as detected on a tumor sample taken within 6 weeks of study entry.
4. At least one measurable site of disease (RECIST Criteria), or other response assessment criteria, as appropriate.
5. Performance status 0,1, 2 or 3 (ECOG).
6. Adequate end organ function.
7. Adequate bone marrow function.
8. Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing.

Exclusion Criteria:

1. Previous treatment with any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
2. Other primary malignancy with < 5 years clinically assessed disease free interval, except basal cell skin cancer, cervical carcinoma in situ, or other neoplasms judged after consultation with the Steering committee to entail a low risk of relapse.
3. Grade III/IV cardiac problems as defined by the New York Heart Association Criteria.
4. Pregnancy, breast-feeding.
5. Severe and/or uncontrolled medical disease.
6. Known brain metastasis.
7. Known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
8. Known diagnosis of human immunodeficiency virus (HIV) infection.
9. Previous treatment with chemotherapy within 4 weeks (6 weeks for nitrosoureas or Mitomycin-C).
10. Previous radiotherapy to ≥ 25 % of the bone marrow.
11. Major surgery within 2 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2002-03; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
tumor response /RecIST criteria) | first 2 months monthly, then every 3 months

SECONDARY OUTCOMES:
SAE and tolerability profile | ongoing basis
OS, DFS | 12 months
effects of the therapy when combined with other treatment modalities i.e. surgery of residual disease. | 12 months
which early predictive factors of tumor response may be of relevance, i.e. conventional pathologic characteristics of tumor and radiological aspects. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- Italy (26):
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Aviano
  - Novartis Investigative Site, Bari
  - Novartis Investigative Site, Bergamo
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Candiolo
  - Novartis Investigative Site, Ferrara
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Livorno
  - Novartis Investigative Site, Meldola
  - Novartis Investigative Site, Messina
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Monserrato
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Nola
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Perugia
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Ravenna
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Rozzano
  - Novartis Investigative Site, Sassari
  - Novartis Investigative Site, Torino
  - Novartis Investigative Site, Verona